CLINICAL TRIAL: NCT02696291
Title: Randomized, Double-blind, Placebo-controlled, Multiple Ascending Dose Study to Determine the Safety, Tolerability and Pharmacokinetics of UV-4B Solution Administered Orally in Healthy Subjects
Brief Title: Safety and Pharmacokinetics of UV-4B Solution Administered Orally as Multiple Ascending Doses to Healthy Subjects
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Product development halted for business reasons.
Sponsor: Emergent BioSolutions (Industry)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DMID 15-0062; HHSN272201100030C (Other Grant/Funding Number: NIAID); 8311-270 (Other: Covance)
Record Dates: First submitted 2016-02-22; First posted 2016-03-02 (Estimated); Results first posted 2018-03-16 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2024-03

CONDITIONS: Viral Infection
Keywords: Dengue; Arbovirus Infections; Flaviviridae Infections; Flavivirus Infections; Hemorrhagic Fevers, Viral; RNA Virus Infections; Virus Diseases; Pharmaceutical Solutions; Pharmacologic Actions; Therapeutic Uses
MeSH Terms: conditions — Virus Diseases; Dengue; Arbovirus Infections; Flaviviridae Infections; Flavivirus Infections; Hemorrhagic Fevers, Viral; RNA Virus Infections | interventions — Solutions

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Cohort 1 - 30 mg (Experimental): Subjects receiving UV-4B 30 mg oral solution or placebo
  Interventions: Drug: UV-4B 30 mg oral solution; Drug: Placebo
- Cohort 2 - 75 mg (Experimental): Subjects receiving UV-4B 75 mg oral solution or placebo
  Interventions: Drug: UV-4B 75 mg oral solution; Drug: Placebo
- Cohort 3 - 150 mg (Experimental): Subjects receiving UV-4B 150 mg oral solution or placebo
  Interventions: Drug: UV-4B 150 mg oral solution; Drug: Placebo
- Cohort 4 - X mg (dose to be determined) (Experimental): Subjects receiving UV-4B X mg (dose to be determined) oral solution or placebo
  Interventions: Drug: UV-4B X mg (dose to be determined) oral solution; Drug: Placebo
- Cohort 5 - Y mg (dose to be determined) (Experimental): Subjects receiving UV-4B Y mg (dose to be determined) oral solution or placebo
  Interventions: Drug: UV-4B Y mg (dose to be determined) oral solution; Drug: Placebo

INTERVENTIONS:
Drug: UV-4B 30 mg oral solution — UV-4B 30 mg oral solution administered TID (every 8 ± 0.5 hours) for 7 days
  Arms: Cohort 1 - 30 mg
Drug: UV-4B 75 mg oral solution — UV-4B 75 mg oral solution administered TID (every 8 ± 0.5 hours) for 7 days
  Arms: Cohort 2 - 75 mg
Drug: UV-4B 150 mg oral solution — UV-4B 150 mg oral solution administered TID (every 8 ± 0.5 hours) for 7 days
  Arms: Cohort 3 - 150 mg
Drug: UV-4B X mg (dose to be determined) oral solution — UV-4B X mg (dose to be determined) oral solution administered TID (every 8 ± 0.5 hours) for 7 days
  Arms: Cohort 4 - X mg (dose to be determined)
Drug: UV-4B Y mg (dose to be determined) oral solution — UV-4B Y mg (dose to be determined) oral solution administered TID (every 8 ± 0.5 hours) for 7 days
  Arms: Cohort 5 - Y mg (dose to be determined)
Drug: Placebo — Placebo oral solution administered TID (every 8 ± 0.5 hours) for 7 days

SUMMARY:
The purpose of this study is to evaluate the safety and pharmacokinetics of UV-4B oral solution when administered to healthy subjects three times a day (TID) for 7 days.

DETAILED DESCRIPTION:
This is a phase 1, randomized, double-blind, placebo-controlled multiple-ascending dose study to evaluate the safety and pharmacokinetics of UV-4B oral solution when administered to healthy subjects TID for 7 days. Three cohorts of 8 subjects each (6 active, 2 placebo) are planned and up to 2 additional cohorts may be added pending safety review of the initial cohorts. Safety review will occur after each cohort. Safety is evaluated through Day 15 on the basis of adverse event (AE) monitoring, clinical laboratory testing (hematology, serum chemistry, coagulation, urinalysis), vital signs, physical examinations (PE), electrocardiograms (ECG), and fecal occult blood testing. Blood samples are collected at specified intervals up to Day 10 for pharmacokinetic assessment.

ELIGIBILITY:
Inclusion Criteria:

* Nonsmoking, healthy male or female subject aged 18 to 45 years, inclusive.
* Female subject is not pregnant and not lactating.
* (Female subjects only who are not postmenopausal or sterile) agreement to use hormonal contraception OR intrauterine device PLUS barrier contraception (condom or occlusive cap such as a diaphragm or surgical vault cap) AND spermicidal foam/gel/cream/suppository starting at least 14 days before the first dose and continuing for at least 3 months after the last dose.
* (Male subjects only) agreement to use barrier contraception during sexual intercourse and to also refrain from sperm donation from the first day of dosing until 3 months after the last dose of the study product.
* Body weight within 60 to 90 kg, inclusive, and body mass index between 18 to 32 kg/m², inclusive.
* Agreement to avoid strenuous exercise starting 4 days before the start of dosing through the period of confinement in the clinical unit and for at least 96 hours before the follow-up visits.

Exclusion Criteria:

* History of allergy to drugs in the iminosugar class.
* Treatment with any investigational products or therapies within 30 days (or 5 half-lives, whichever is greater) before the first day of dosing.
* Current or past history of disease/dysfunction of the pulmonary, cardiovascular, endocrine, hematologic, neurological, immune, gastrointestinal genitourinary, or other body system.
* Abnormalities on physical examination suggestive of conditions that may pose an increased risk to the subject; abnormal electrocardiogram results (excluding benign conditions); and Grade 1 or higher abnormalities in vital signs at screening and Grade 2 or higher abnormalities in vital signs at check-in based on a modified version of the FDA Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials.
* Clinical laboratory tests outside the normal range at screening and Grade 2 or higher at check-in to the clinical unit.
* Creatinine clearance < 90 mL/min (based on Cockcroft-Gault equation).
* Proteinuria greater than or equal to 1+.
* Any known or expected risk of bleeding.
* Scheduled surgical procedure during study participation.
* History of alcohol and/or drug abuse within 1 year prior to dosing and/or a positive urine drug screen for substances of abuse at screening or check-in. Urine alcohol above 50 mg/dL.
* Plasma or blood donation within 30 days before the first day of dosing or intention to donate within 30 days after the final day of dosing.
* Treatment with any medication, either prescription or nonprescription, including dietary supplements or herbal medications, within 14 days before dosing (within 30 days before dosing for hepatic or renal clearance-altering agents) and is unable to refrain from any medication during the study period. Exceptions are acetaminophen (not more than 2 g/day), vitamin products at recommended daily doses or hormonal birth control.
* Positive serology test for HIV antibodies, hepatitis B surface antigen, or hepatitis C virus antibody at screening.
* History of relevant food allergies (ie, eggs or other components of standard clinic meals) or unwilling to comply with diet restrictions.
* Psychological and/or emotional problems which would render the informed consent invalid, or limit the ability of the subject to comply with the study requirements;
* Concurrent enrollment in any other clinical trial within 30 days.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 7 (Actual)
Dates: Start 2016-05-27 (Actual); Primary Completion 2017-03-02 (Actual); Study Completion 2017-03-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Babinchak, MD, Study Director — Emergent BioSolutions
Locations (2):
- United States (2):
  - Clinical Research Unit, Dallas, Texas
  - Clinical Research Unit, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: For information on dengue fever — https://www.niaid.nih.gov/diseases-conditions/dengue-fever

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Healthy subjects were recruited from a phase 1 clinical research unit. Recruitment was initiated on 27 May 2016 and the last subject completed the final study visit for Cohort 1 on 02 March 2017.
Groups:
- Cohort 1 - 30 mg UV-4B: Subjects receiving UV-4B 30 mg oral solution TID (every 8 ± 0.5 hours) for 7 days
- Cohort 1 - Placebo: Subjects receiving placebo TID (every 8 ± 0.5 hours) for 7 days
Period: Overall Study
Arm/Group | Cohort 1 - 30 mg UV-4B | Cohort 1 - Placebo
Started | 5 | 2
Completed | 5 | 2
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 - 30 mg UV-4B | Cohort 1 - Placebo | Total
Number analyzed (Participants) | 5 | 2 | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.2 (8.3) | 41.5 (4.9) | 34.1 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 5
  Male | 2 | 0 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 3
  Not Hispanic or Latino | 3 | 1 | 4
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 4 | 2 | 6
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 26.0 (1.0) | 28.4 (2.3) | 26.7 (1.7)

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Reporting Treatment-emergent Adverse Events (TEAEs) by Group
Description: The incidence of TEAEs spontaneously reported by subjects or elicited during examination is reported by dose group. Subjects having multiple TEAEs are counted only once.
Time Frame: From the time of first dosing on Day 1 through the Day 15 final follow-up visit
Population: Safety Population: all subjects who received at least one dose of study product or placebo.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 - 30 mg UV-4B | Cohort 1 - Placebo
Number analyzed (Participants) | 5 | 2
Participants | 5 | 2

2. Primary Outcome: Number of Subjects Reporting Serious Adverse Events (SAEs) by Group
Description: The incidence of SAEs spontaneously reported by subjects or elicited during examination is reported by dose group. Subjects having multiple SAEs are counted only once.
Time Frame: From the time of first dosing on Day 1 through the Day 15 final follow-up visit
Population: Safety Population: all subjects who received at least one dose of study product or placebo.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 - 30 mg UV-4B | Cohort 1 - Placebo
Number analyzed (Participants) | 5 | 2
Participants | 1 | 0

3. Primary Outcome: Number of Subjects With Clinical Laboratory Abnormalities of Toxicity Grade 1 or Higher by Group
Description: Clinical laboratory abnormalities are presented as the total of Grade 1 (mild) through Grade 4 (potentially life-threatening) abnormalities according to criteria adapted from the Food and Drug Administration (FDA) Guidance for Industry, Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials (September 2007) and the Division of Microbiology and Infectious Diseases (DMID) Adult Toxicity Table (November 2007). Within each parameter, subjects having multiple abnormalities are counted only once.
Time Frame: From the time of first dosing on Day 1 through the Day 15 final follow-up visit
Population: Safety Population: all subjects who received at least one dose of study product or placebo.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 - 30 mg UV-4B | Cohort 1 - Placebo
Number analyzed (Participants) | 5 | 2
Participants
  Any ≥ Grade 1 result | 5 | 2
  ≥ Grade 1 activated partial thromboplastin time | 1 | 0
  ≥ Grade 1 hemoglobin decreased | 5 | 2
  ≥ Grade 1 leukocytes decreased | 1 | 0
  ≥ Grade 1 magnesium decreased | 0 | 1
  ≥ Grade 1 prothrombin time increased | 4 | 1
  ≥ Grade 1 sodium decreased | 1 | 0
  ≥ Grade 1 urine erythrocytes (present) | 4 | 2

4. Secondary Outcome: Number of Subjects With Outlying Vital Sign Results by Group
Description: Vital signs of blood pressure (BP), pulse, respiratory rate, and oral temperature were taken after being supine for 10 minutes. Orthostatic vital signs (BP, pulse) were taken after 2 minutes standing. Vital sign results are presented as the number of subjects having Grade 1 (mild) through Grade 4 (potentially life-threatening) abnormalities according to criteria adapted from the FDA Guidance for Industry, Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials (September 2007), or having abnormal orthostatic change (standing minus supine result). Within each parameter, subjects having multiple abnormalities are counted only once.
Time Frame: From the time of first dosing on Day 1 through the Day 15 final follow-up visit
Population: Safety Population: all subjects who received at least one dose of study product or placebo.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 - 30 mg UV-4B | Cohort 1 - Placebo
Number analyzed (Participants) | 5 | 2
Participants
  Any ≥ Grade 1 result | 5 | 2
  ≥ Grade 1 supine systolic BP ≤ 89 mmHg | 1 | 0
  ≥ Grade 1 supine pulse ≤ 50 bpm (if baseline ≤ 60) | 1 | 0
  ≥ Grade 1 supine pulse ≤ 54 bpm (if baseline > 60) | 1 | 0
  ≥ Grade 1 supine pulse ≥ 101 bpm | 0 | 1
  ≥ Grade 1 respiratory rate ≥ 17 breaths/min | 2 | 1
  Any orthostatic change | 5 | 2
  Orthostatic change in diastolic BP ≤ -10 mmHg | 1 | 1
  Orthostatic change in pulse > 30 bpm | 5 | 1

5. Secondary Outcome: Number of Subjects With 12-lead Electrocardiogram (ECG) Abnormalities Postdose by Group
Description: ECGs (ventricular heart rate, wave intervals - PR, QRS, QT, QTcF) were recorded in a supine position (for at least 10 minutes). Baseline was calculated from the average of the triplicate ECGs on Day 1 predose. Within each parameter, subjects having multiple abnormalities are counted only once.
Time Frame: From the time of first dosing on Day 1 through the Day 15 final follow-up visit
Population: Safety Population: all subjects who received at least one dose of study product or placebo.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 - 30 mg UV-4B | Cohort 1 - Placebo
Number analyzed (Participants) | 5 | 2
Participants
  Any ECG abnormality | 2 | 0
  PR > 220 ms | 2 | 0

6. Secondary Outcome: Maximum Plasma Concentration (Cmax)
Description: Plasma concentrations of UV-4 are determined by means of high performance liquid chromatography/tandem mass spectrometric assay. Values of Cmax are derived from individual subject plasma concentration-time data. Blood collected at 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 5, 6, and 8 hrs after the first dose on Day 1; and at 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 5, 6, 8, 10, 12, and 14 hrs after the final dose on Day 7.
Time Frame: Day 1, Day 7
Population: Pharmacokinetic Population: all subjects who received study product, had measurable values, and completed scheduled postdose pharmacokinetic measurements without protocol deviations or events thought to significantly affect the pharmacokinetics of the drug.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Cohort 1 - 30 mg UV-4B
Number analyzed (Participants) | 5
ng/mL
  Day 1 Cmax | 291 (15.8)
  Day 7 Cmax | 285 (5.1)

7. Secondary Outcome: Time of Maximum Plasma Concentration (Tmax)
Description: Plasma concentrations of UV-4 are determined by means of high performance liquid chromatography/tandem mass spectrometric assay. Values of tmax are derived from individual subject plasma concentration-time data. Blood collected at 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 5, 6, and 8 hrs after the first dose on Day 1; and at 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 5, 6, 8, 10, 12, and 14 hrs after the final dose on Day 7.
Time Frame: Day 1, Day 7
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: h
Arm/Group | Cohort 1 - 30 mg UV-4B
Number analyzed (Participants) | 5
h
  Day 1 tmax | 0.7 (0.2)
  Day 7 tmax | 1.0 (0.4)

8. Secondary Outcome: Area Under the Concentration-time Curve From Time Zero (Predose) to Time of the Last Quantifiable Concentration After the Last Dose [AUC(0-last)]
Description: Plasma concentrations of UV-4 are determined by means of high performance liquid chromatography/tandem mass spectrometric assay. Values of AUC(0-last) are derived from individual subject plasma concentration-time data, calculated using the linear trapezoidal rule for increasing concentrations and the logarithmic rule for decreasing concentrations. Blood collected at 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 5, 6, 8, 10, 12, and 14 hrs after the final dose on Day 7.
Time Frame: Day 7
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Cohort 1 - 30 mg UV-4B
Number analyzed (Participants) | 5
ng*hr/mL | 1800 (14.2)

9. Secondary Outcome: Total Daily Exposure at Steady State: Area Under the Concentration-time Curve From Time Zero (Predose) Until 24 Hours After the Last Dose [AUC(0-24)]
Description: Plasma concentrations of UV-4 are determined by means of high performance liquid chromatography/tandem mass spectrometric assay. Values of AUC(0-24) are derived from individual subject plasma concentration-time data, calculated as AUC(0-8) x 3 (Day 7 last dose only). Blood collected at 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 5, 6, 8, 10, 12, and 14 hrs after the final dose on Day 7.
Time Frame: Day 7
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Cohort 1 - 30 mg UV-4B
Number analyzed (Participants) | 5
ng*hr/mL | 3810 (3.7)

10. Secondary Outcome: Area Under the Concentration-time Curve From Time Zero (Predose) Until 8 Hours After the Final Dose [AUC(0-8)]
Description: Plasma concentrations of UV-4 are determined by means of high performance liquid chromatography/tandem mass spectrometric assay. Values of AUC(0-8) are derived from individual subject plasma concentration-time data, calculated using the linear trapezoidal rule for increasing concentrations and the logarithmic rule for decreasing concentrations. Blood collected at 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 5, 6, and 8 hrs after the first dose on Day 1; and at 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 5, 6, 8, 10, 12, and 14 hrs after the final dose on Day 7.
Time Frame: Day 1, Day 7
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Cohort 1 - 30 mg UV-4B
Number analyzed (Participants) | 5
ng*hr/mL
  Day 1 AUC(0-8) | 965 (8.7)
  Day 7 AUC(0-8) | 1270 (3.7)

11. Secondary Outcome: Apparent Systemic Clearance (CL/F) at Steady State
Description: Plasma concentrations of UV-4 are determined by means of high performance liquid chromatography/tandem mass spectrometric assay. Values of CL/F are derived from individual subject plasma concentration-time data, calculated as dose (free-base equivalent) divided by AUC(0-8). Blood collected at 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 5, 6, 8, 10, 12, and 14 hrs after the final dose on Day 7.
Time Frame: Day 7
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/h
Arm/Group | Cohort 1 - 30 mg UV-4B
Number analyzed (Participants) | 5
L/h | 23.6 (3.7)

12. Secondary Outcome: Apparent Volume of Distribution of UV-4 During the Terminal Phase (Vz/F) After Multiple Doses
Description: Plasma concentrations of UV-4 are determined by means of high performance liquid chromatography/tandem mass spectrometric assay. Values of Vz/F are derived from individual subject plasma concentration-time data, calculated as CL/F divided by λz. Blood collected at 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 5, 6, 8, 10, 12, and 14 hrs after the final dose on Day 7.
Time Frame: Day 7
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L
Arm/Group | Cohort 1 - 30 mg UV-4B
Number analyzed (Participants) | 5
L | 246 (30.6)

13. Secondary Outcome: Apparent Terminal Half Life (t1/2)
Description: Plasma concentrations of UV-4 are determined by means of high performance liquid chromatography/tandem mass spectrometric assay. Values of t1/2 are derived from individual subject plasma concentration-time data, calculated as ln2/λz. Blood collected at 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 5, 6, 8, 10, 12, and 14 hrs after the final dose on Day 7.
Time Frame: Day 7
Population: as for outcome 6
Measure: Median (Full Range); unit: h
Arm/Group | Cohort 1 - 30 mg UV-4B
Number analyzed (Participants) | 5
h | 8.1 [4.1 to 9.0]

14. Secondary Outcome: Accumulation Ratio (AR)
Description: Accumulation Ratio (AR) Day 1/Day 7
Time Frame: Day 7
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Cohort 1 - 30 mg UV-4B
Number analyzed (Participants) | 5
Ratio | 1.3 (5.8)

ADVERSE EVENTS:
Time Frame: Up to Day 15.
Description: On-treatment SAEs and non-serious AEs were collected from the start of investigational product until Day 15.
Arm/Group | Cohort 1 - 30 mg UV-4B | Cohort 1 - Placebo
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/2
Serious Adverse Events (participants affected / at risk) | 1/5 | 0/2
Other Adverse Events (participants affected / at risk) | 5/5 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 - 30 mg UV-4B (N=5) | Cohort 1 - Placebo (N=2)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Cohort 1 - 30 mg UV-4B (N=5) | Cohort 1 - Placebo (N=2)
Atrioventricular block first degree (Cardiac disorders) | 1 (1) | 0 (0)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Flatulence (Gastrointestinal disorders) | 2 (2) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Epigastric discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gingival bleeding (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vessel puncture site haematoma (General disorders) | 1 (1) | 1 (1)
Vessel puncture site pain (General disorders) | 1 (1) | 1 (1)
Vessel puncture site haemorrhage (General disorders) | 0 (0) | 1 (1)
Haemoglobin decreased (Investigations) | 5 (5) | 2 (2)
Prothrombin time prolonged (Investigations) | 4 (4) | 1 (1)
Activated partial thromboplastin time (Investigations) | 1 (1) | 0 (0)
White blood cell count decreased (Investigations) | 1 (1) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 3 (3) | 2 (2)
Testis discomfort (Reproductive system and breast disorders) | 1/2 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Study was terminated after Cohort 1. While no analysis was performed for change from baseline for physical exam (PE, a secondary endpoint), any change from baseline PE was reported/analyzed as an AE. AUC0-inf (secondary endpoint) was not calculated.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2017-01-10): https://cdn.clinicaltrials.gov/large-docs/91/NCT02696291/Prot_001.pdf
  • Statistical Analysis Plan (2017-05-31): https://cdn.clinicaltrials.gov/large-docs/91/NCT02696291/SAP_000.pdf